CLINICAL TRIAL: NCT02815696
Title: MRI Analysis of Glycosaminoglycan Modifications Inside the Intervertebral Disk After Distraction and Posterior Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tamas Illes, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-DGemric
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Lumbar Spine Instability
Keywords: MRI T2 weighted; intervertebral disc; glycosaminoglycans
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lumbar spine segmental instability (Experimental): Patients with a segmental instability of the lumbar spine having undergone surgery. Lumbar spine instability diagnosis is based on imaging (Magnetic resonance imaging, standard radiography, and EOS imaging). Surgical treatment is indicated if the pain is relieved by wearing a brace during at least three months.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Specific MRI sequences (delayed gadolinium-enhanced magnetic resonance imaging of cartilage -dGEMRIC) performed before the surgery, 6 months and 1 year after surgery will allow to measure the following parameters: disc height, total lumbar spine lenght, GAGs concentration.

SUMMARY:
Degenerative disc disease (DDD) is the primary cause of low back pain. The most important factor in the development of DDD is the vertical load force on the disc, increasing the hydrostatic pressure and facilitating discs degenerations. One of the most common conditions accompanying DDD is segmental instability of the spine. The pathogenesis evolves in three phases characterized by a progressive disc dehydration and loss of the disc height.

This phenomenon can be observed in magnetic resonance imaging (T2 weighted MRI) as a decrease of the water signal inside the intervertebral disc. It is considered as an indirect sign of the alteration of the composition (including glycosaminoglycans) and the structure of the intervertebral disk with, as consequence, a modification of the spine biomechanics. Animal studies showed that disc regeneration could be enhanced by a decrease of the hydrostatic pressure. This could be observed as a signal increase on T2 weighted MRI.

Recent quantitative MRI sequences now allow the quantification of glycosaminoglycans (GAG) concentration inside the cartilage and in the intervertebral disc.

The actual surgical trends are in favor of an anterior (intersomatic) vertebrak fusion, associated or not with a posterior fusion. These technics sacrifice the intervertebral disc and change the spine biomechanics.

Based on a pilot study, the investigators believe that the conservation and even a regeneration of the intervertebral disc is possible and allows the preservation of the spine biomechanics.

The purpose of the study is to analyze the relations between specific MRI signals, the GAGs concentration, and the functional outcome before and after the surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with segmental instability of the lumbar spine
* Patient with planned surgery

Exclusion Criteria:

* clinical and iconographic signs of neurological compression
* intervertebral disc completely degenerated
* infection
* spondylolisthesis (superior to grade I)
* fracture
* neoplasia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Gycosaminoglycan (GAG) concentration of the intervertebral disk | Baseline: before surgery
  GAG concentration is estimated using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Gycosaminoglycan (GAG) concentration of the intervertebral disk | Six months after surgery
  GAG concentration is estimated using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Gycosaminoglycan (GAG) concentration of the intervertebral disk | 1 year after surgery
  GAG concentration is estimated using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique

SECONDARY OUTCOMES:
Disc height | Baseline: before surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Disc height | Six months after surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Disc height | 1 year after surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Total lumbar spine length | Baseline: before surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Total lumbar spine length | Six months after surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Total lumbar spine length | 1 year after surgery
  Will be measured using the delayed gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) technique
Lumbar lordosis angle | Baseline: before surgery
  Will be measured by the EOS imaging system.
Lumbar lordosis angle | Six months after surgery
  Will be measured by the EOS imaging system.
Lumbar lordosis angle | 1 year after surgery
  Will be measured by the EOS imaging system.
Oswestry Disability Index (ODI) | Baseline: before surgery
  Estimation of the functional state of the patient by the Oswestry Disability questionnaire.
Oswestry Disability Index (ODI) | Six months after surgery
  Estimation of the functional state of the patient by the Oswestry Disability questionnaire.
Oswestry Disability Index (ODI) | 1 year after surgery
  Estimation of the functional state of the patient by the Oswestry Disability questionnaire.
SF-36 | Baseline: before surgery
  Estimation of the functional state of the patient by the SF-36 questionnaire relative to the quality of life.
SF-36 | Six months after surgery
  Estimation of the functional state of the patient by the SF-36 questionnaire relative to the quality of life.
SF-36 | 1 year after surgery
  Estimation of the functional state of the patient by the SF-36 questionnaire relative to the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Illes, MD, Principal Investigator — CHU Brugmann; Dinh Qui Du PHAN, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Singh V, Datta S, Cohen SP, Hirsch JA; American Society of Interventional Pain Physicians. Comprehensive review of epidemiology, scope, and impact of spinal pain. Pain Physician. 2009 Jul-Aug;12(4):E35-70. PMID 19668291
- [Background] Iatridis JC, MacLean JJ, Roughley PJ, Alini M. Effects of mechanical loading on intervertebral disc metabolism in vivo. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2(0 2):41-6. doi: 10.2106/JBJS.E.01407. PMID 16595442
- [Background] Haughton V. The "Dehydrated" Lumbar Intervertebral Disk on MR, its Anatomy, Biochemistry and Biomechanics. Neuroradiol J. 2011 Aug 31;24(4):564-9. doi: 10.1177/197140091102400412. Epub 2011 Sep 2. PMID 24059714
- [Background] Kroeber M, Unglaub F, Guehring T, Nerlich A, Hadi T, Lotz J, Carstens C. Effects of controlled dynamic disc distraction on degenerated intervertebral discs: an in vivo study on the rabbit lumbar spine model. Spine (Phila Pa 1976). 2005 Jan 15;30(2):181-7. doi: 10.1097/01.brs.0000150487.17562.b1. PMID 15644753
- [Background] Gray ML. Toward imaging biomarkers for glycosaminoglycans. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1(Suppl 1):44-9. doi: 10.2106/JBJS.H.01498. PMID 19182023